CLINICAL TRIAL: NCT06660511
Title: Exploratory Study on the Safety and Efficacy of Disitamab Vedotin in Combination with Anlotinib Hydrochloride for the Treatment of HER-2-expressing Recurrent Platinum-resistant Ovarian Cancer.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jingjing Wang, associate chief physician, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYEC2024-0343
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer Recurrent
Keywords: Ovarian Cancer Recurrent
MeSH Terms: interventions — disitamab vedotin; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): The dose of Disitamab Vedotin(RC48) is 2.0 mg/kg iv q2w d1; The dose of Anlotinib Hydrochloride Capsules is 10mg po qd (recommended to be taken before meals and at the same time every day), taken orally continuously for 2 weeks and stopped for 1 week, with a treatment cycle of 21 days.
  Interventions: Drug: Disitamab Vedotin in Combination With Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Disitamab Vedotin in Combination With Anlotinib Hydrochloride — The dose of Disitamab Vedotin(RC48) is 2.0 mg/kg iv q2w d1; The dose of Anlotinib Hydrochloride Capsules is 10mg po qd (recommended to be taken before meals and at the same time every day), taken orally continuously for 2 weeks and stopped for 1 week, with a treatment cycle of 21 days.
  Main research endpoint: Objective response rate (ORR)
  Secondary study endpoint:
  1. Progression free survival (PFS)
  2. Overall survival (OS)
  3. Disease Control Rate (DCR)
  4. Objective Duration of Response (DoR)
  Other Names: RC48 combined with Anlotinib Hydrochloride; RC48 combined with AL3818; RC48 combined with Anlotinib

SUMMARY:
Ovarian cancer is one of the three major malignant tumors of the female reproductive system. Even if newly diagnosed ovarian cancer patients undergo ideal tumor cell reduction surgery and postoperative chemotherapy, 70% to 80% of ovarian cancer patients still experience recurrence. According to the length of PFI (platinum free interval), recurrent ovarian cancer (ROC) can be classified into platinum resistant ROC (<6 months) and platinum sensitive ROC (>6 months). There is currently no optimal treatment plan for platinum resistant ovarian cancer (PROC), and the prognosis for patients is poor. The guidelines recommend non platinum monotherapy chemotherapy for patients with PROC, but non platinum monotherapy has a low objective response rate (ORR) (<20%), progression free survival (PFS) (<4 months), and overall survival (OS,<12 months), with significant adverse reactions and affecting quality of life. Therefore, PROC patients urgently need new and better treatment options.

Antibody conjugated drugs (ADCs) have made breakthrough therapeutic progress in multiple tumor types, and currently ADCs have been approved by the FDA for the treatment of cervical cancer and ovarian cancer. HER2 (Human Epidermal Growth Factor Receptor 2) is a member of the epidermal growth factor receptor (EGFR) family, also known as the tyrosine protein kinase receptor. Research has shown that HER2 expression is associated with poor prognosis in ovarian cancer, and patients with HER2 positive expression have a worse prognosis. Vidiximab (RC48) is a novel HER2 antibody conjugate drug that received Breakthrough Therapy Design from the US Food and Drug Administration (FDA) in April 2020. Preclinical studies of ovarian cancer have shown that vediximab exhibits effective cytotoxicity against HER2 expressing ovarian tumor cell lines. Meanwhile, the registration study of RC48 for gynecological tumors is underway, and its latest data was reported at the 2024 European Congress of Gynecological Oncology (ESGO), which showed that in patients with recurrent or metastatic cervical cancer, the ORR of RC48 monotherapy was 36.4%, the median PFS was 4.37 months, and the 1-year OS was 66%. Compared to other chemotherapy drugs, it also has significant advantages in terms of toxic side effects, with severity mostly ranging from grade 1-2. Symptomatic treatment can achieve complete recovery or relief.

Anti angiogenic drugs, including anti vascular endothelial growth factor (VEGF) antibodies and multi-target tyrosine kinase inhibitors (TKIs), are considered potential targets for treating platinum resistant/refractory ovarian diseases . Anlotinib is a novel oral multi-target tyrosine kinase inhibitor (TKIs) . Monotherapy for PROC has achieved initial efficacy, with an ORR of 31.2%, a median PFS of 5.3 months, and a 12-month OS rate of 90.9%. In terms of safety, most of the toxic side effects are grade 1-2.

Good progress has been made in preclinical and clinical trials of ADC in combination with other anti-cancer drugs, including chemotherapy, molecular targeted drugs, anti angiogenic drugs, and immunotherapy. Among them, anti angiogenic drugs may promote the penetration and exposure of ADC to tumor cells, playing a mutually reinforcing role. Research on the combination of RC48 and anlotinib is also actively underway in other tumor types.

In summary, this study creatively conducted exploratory research in clinical PROC patients based on the different expression levels of the molecular target HER2, and adopted targeted medication according to the molecular target. At the same time, in terms of combination therapy, low toxicity and high efficiency, different toxic side reaction spectra, different mechanisms of action, and synergistic effects of dual anti-tumor drugs were selected for combination therapy. Based on the above evidence, an exploratory study was conducted on the safety and efficacy of vediximab combined with anlotinib in the treatment of HER-2 expressing recurrent platinum resistant ovarian cancer, aiming to explore the efficacy of vediximab combined with anlotinib in PROC patients, in order to further improve the remission rate and quality of life of patients while prolonging their survival.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed an informed consent form, and showed good compliance;
2. Age ≥ 18 years old when signing the informed consent form;
3. Epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer diagnosed by organizational or cellular pathology;
4. The subjects can provide tumor primary or metastatic site specimens for HER2 detection (paraffin blocks, paraffin embedded sections, or fresh tissue sections are all acceptable), and the immunohistochemical (IHC) test results show HER2 expression: IHC 1+, 2+, or 3+; 4) ECOG PS: 0-1 point;
5. Expected survival period>12 weeks;
6. Adequate heart, bone marrow, liver, and kidney function (based on normal values at the research center);
7. At least one measurable lesion defined in RECIST version 1.1;
8. Women of childbearing age must meet one of the following conditions:

   * Surgical sterilization has been performed; ② Menopausal individuals who have stopped menstruating for at least one year; ③ Having the ability to conceive requires meeting the following conditions:; The serum pregnancy test result before the first medication is negative and must be a non lactating subject; During the entire study period, it was agreed to use a recognized method of contraception (such as oral contraception, injection contraception, or implanted barrier contraception, spermicides and condoms, or intrauterine devices), and the contraceptive method remained unchanged throughout the study period.

Exclusion criteria：

1. Previously received ADC drugs for HER2 treatment or similar TKI small molecule anti angiogenic drugs such as anlotinib hydrochloride;
2. Subjects with primary platinum refractory diseases;
3. Patients with untreated central nervous system metastases (including new and progressive brain metastases), a history of leptomeningeal metastases or malignant meningitis;
4. Individuals with symptoms and signs of intestinal obstruction and requiring parenteral nutrition and fluid replacement;
5. Patients with any signs of bleeding or history of bleeding, regardless of the severity: patients who have experienced any bleeding or bleeding events ≥ CTCAE grade 3 within the 4 weeks prior to the first dose; Or there may be unhealed wounds, fractures, active ulcers in the stomach and duodenum, ulcerative colitis and other digestive diseases.
6. Within 6 months, there have been incidents of arterial/venous thrombosis, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; (Individuals with a tendency towards thrombosis or undergoing anticoagulant therapy are allowed to use prophylactic anticoagulant therapy)
7. Serious cardiovascular and cerebrovascular diseases or discomfort, including but not limited to the following diseases:

   * Diagnosed history of heart failure or systolic dysfunction (LVEF<50%)
   * High risk uncontrolled arrhythmia
   * Angina pectoris, acute myocardial infarction
   * Clinically significant heart valve disease
   * Poor control of hypertension (systolic blood pressure>180 mmHg and/or diastolic blood pressure>100 mmHg)
8. The toxicity caused by previous anti-tumor treatments has not yet recovered to CTCAE (version 5.0) grade 0-1 (excluding 2nd degree hair loss);
9. Individuals who have undergone major surgery within 4 weeks prior to their first medication and have not fully recovered, or are expected to undergo surgical treatment;
10. Patients with other malignant tumors within 3 years prior to the first use of medication, excluding papillary thyroid carcinoma, basal cell or squamous cell carcinoma that have been adequately treated and have no evidence of disease recurrence, as well as other in situ cancers that have been adequately treated and have no evidence of disease recurrence (including but not limited to cervical primary cancer, ductal carcinoma in situ of the breast, etc.);
11. Imaging (CT or MRI) shows that the tumor has invaded important blood vessels or is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies, as determined by the researcher;
12. Patients with clinical symptoms of pleural effusion, pericardial effusion, or ascites who require repeated puncture and drainage, or those who have received treatment within the previous month for the purpose of drainage;
13. Individuals with a known history of allergies to the components of this medication regimen;
14. Pregnant and lactating female patients;
15. Suffering from serious accompanying diseases or other comorbidities that may interfere with planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR): The proportion of subjects whose best overall response rate (BOR) is evaluated as complete response (CR) or partial response (PR) according to RECIST 1.1 criteria. | From the initial use of medication until disease progression, death, initiation of new anti-tumor treatment, loss to follow-up, withdrawal of informed consent, and completion of the study, evaluation is conducted for 2 years.

SECONDARY OUTCOMES:
From the date of enrollment to the date of the first recorded tumor progression (assessed according to RECIST 1.1 criteria, regardless of whether treatment is continued or not) or the date of death from any cause for the subjects. | From the initial use of medication until disease progression, death, initiation of new anti-tumor treatment, loss to follow-up, withdrawal of informed consent, and completion of the study, evaluation is conducted for 2 years.
  Progression free survival (PFS): defined as the period from enrollment to the date of the first recorded tumor progression (assessed according to RECIST 1.1 criteria, regardless of whether treatment is continued or not) or the date of death from any cause, whichever occurs first.
Overall survival (OS): defined as the time between enrollment and death of the subject due to various reasons, and calculated based on the intention to treat population (ITT). | From the initial use of medication until disease progression, death, initiation of new anti-tumor treatment, loss to follow-up, withdrawal of informed consent, and completion of the study, evaluation is conducted for 2 years.
Disease Control Rate (DCR): The proportion of subjects with the best overall response (BOR) evaluated according to RECIST 1.1 criteria as complete response (CR), partial response (PR), and disease stability (SD). | From the initial use of medication until disease progression, death, initiation of new anti-tumor treatment, loss to follow-up, withdrawal of informed consent, and completion of the study, evaluation is conducted for 2 years.
Duration of Response (DoR): defined as the period from the first recorded tumor response (assessed according to RECIST 1.1 criteria) to the first recorded objective tumor progression (assessed according to RECIST 1.1 criteria) or death from any cause. | From the initial use of medication until disease progression, death, initiation of new anti-tumor treatment, loss to follow-up, withdrawal of informed consent, and completion of the study, evaluation is conducted for 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Second Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided